CLINICAL TRIAL: NCT03858179
Title: Effects of Photobiomodulation Therapy in Strength Training and Detraining in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1781602
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Muscle Strength
Keywords: Photobiomodulation Therapy; Low-level Laser Therapy; Skeletal Muscle Strenght; Strength Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A researcher will program the device (placebo or PMBT) and will be instructed not to inform the volunteers or other researchers as to the type of treatment (PMBT or placebo). Therefore, the researcher responsible for the treatment will be blinded to the type of treatment being administered to the volunteers. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (placebo or PBMT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PBMT + training/ PBMT + detraining (Experimental): PBMT applied before the strength training sessions (12 weeks, 2 times a week) and PBMT applied during the detraining period (4 weeks, 2 times a week).
  Interventions: Device: PBMT
- PBMT + training/ placebo + detraining (Experimental): PBMT applied before the strength training sessions (12 weeks, 2 times a week) and placebo applied during the detraining period (4 weeks, 2 times a week).
  Interventions: Device: PBMT; Device: Placebo
- Placebo + training/ PBMT + detraining (Experimental): Placebo applied before the strength training sessions (12 weeks, 2 times a week) and PBMT applied during the detraining period (4 weeks, 2 times a week).
  Interventions: Device: PBMT; Device: Placebo
- Placebo + training/ placebo + detraining (Placebo Comparator): Placebo applied before the strength training sessions (12 weeks, 2 times a week) and placebo applied during the detraining period (4 weeks, 2 times a week).
  Interventions: Device: Placebo

INTERVENTIONS:
Device: PBMT — PBMT will be applied bilaterally using the direct contact method with light pressure on the skin to 6 sites of the anterior thigh (2 medial, 2 lateral, and 2 central). A 12-diode cluster, with 4 905-nm laser diodes (12.5W peak power for each diode), 4 875-nm LED diodes (17.5 mW mean power for each diode), and 4 640-nm LED diodes (15 mW mean power for each diode), manufactured by Multi Radiance Medical® (Solon, OH, USA), will be used to apply the PBMT. The dose used for applications during the training and/or detraining periods will be 30 Joules (J) per site (180 J per thigh). PBMT will be applied before each workout and during the detraining period, depending on the group to which the volunteers are allocated.
  Arms: PBMT + training/ PBMT + detraining; PBMT + training/ placebo + detraining; Placebo + training/ PBMT + detraining
Device: Placebo — Placebo PBMT will be applied bilaterally using the direct contact method with light pressure on the skin to 6 sites of the anterior thigh (2 medial, 2 lateral, and 2 central). The placebo PBMT will per performed using the dose of 0 J per diode. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (active or placebo). Placebo PBMT will be applied before each workout and during the detraining period, depending on the group to which the volunteers are allocated.
  Arms: PBMT + training/ placebo + detraining; Placebo + training/ PBMT + detraining; Placebo + training/ placebo + detraining

SUMMARY:
In last years it has been demonstrated that photobiomodulation therapy (PBMT) has ergogenic effects, improving muscular performance and accelerating post-exercise recovery. However, many aspects related to these effects and its' clinical applicability remain unknown. Therefore, the aim of this project is to evaluate the ergogenic effects of PBMT in detraining after a strength training protocol.

DETAILED DESCRIPTION:
It will be carried out a randomized, triple-blind, placebo-controlled trial.

Forty-eight volunteers will be randomly allocated to four experimental groups:

1. PBMT before the strength training sessions and PBMT during the detraining period;
2. PBMT before the strength training sessions and placebo during the detraining period;
3. Placebo before the strength training sessions and PBMT during the detraining period;
4. Placebo before the strength training sessions and placebo during the detraining period .

The individuals randomly allocated to the different groups will be subjected to 12 consecutive weeks of dynamic strength training involving leg-press and knee extension exercises in leg-press and leg-extension machines, respectively, 2 times a week.After the 12-week training period, the volunteers will receive the application of PBMT or placebo depending on the group to which they are allocated for 4 weeks (2 times a week) without training.

The data will be collected by a blind assessor. It will be analyzed the muscular strength and the structural properties of quadriceps before starting the study (baseline), at 4, 8, and 12 weeks after starting the training period, and at 4 weeks after completing the training (detraining period), in both lower limbs.

The findings will be tested for their normality using the Shapiro-Wilk test. Parametric data will be expressed as mean and standard deviation and non-parametric data as median and respective upper and lower limits. Parametric data will be analyzed by two-way repeated measures analysis of variance (ANOVA; time versus experimental group) with post-hoc Bonferroni correction. Non-parametric data will be analyzed using the Friedman test and, secondarily, the Wilcoxon signed-rank test. Data will be analyzed in terms of both their absolute values and their relationship to the percentage change based on the values established in the baseline tests. The significance level will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men;
* Aged from 18 to 35 years;
* Complete at least 80% of the study procedures will be included in the study.

Exclusion Criteria:

* History of musculoskeletal injury in the hip and knee regions in the 2 months before the study;
* Become injured during the study;
* Regularly use pharmacological agents and/ or nutritional supplements;
* Signs and symptoms of any neurological, metabolic, inflammatory, pulmonary, oncological, or cardiovascular disease that may limit the execution of high-intensity exercises.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Peak Torque | 16 weeks - 4 weeks after completing the training (detraining period).
  The peak torque will be measured by Maximum Voluntary Contraction (MVC) test.

SECONDARY OUTCOMES:
Peak Torque | 4, 8, and 12 weeks after starting the training period.
  The peak torque will be measured by Maximum Voluntary Contraction (MVC) test.
Muscle strength | 4, 8, and 12 weeks after starting the training period, and at 4 weeks after completing the training (detraining period).
  Muscle strength will be measured by one-repetition maximum (1-RM) test.
Muscle thickness | 4, 8, and 12 weeks after starting the training period, and at 4 weeks after completing the training (detraining period).
  Muscle thickness will be measured by ultrasound imaging.
Muscle fascicle length | 4, 8, and 12 weeks after starting the training period, and at 4 weeks after completing the training (detraining period).
  Muscle fascicle length will be measured by ultrasound imaging.
Muscle fiber pennation angle | 4, 8, and 12 weeks after starting the training period, and at 4 weeks after completing the training (detraining period).
  Muscle fiber pennation angle will be measured by ultrasound imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Cesar Pinto Leal Junior, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Laboratory of Phototherapy and Innovative Technologies in Health, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request addressed to the principal investigator.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] de Paiva PRV, Tomazoni SS, Machado CDSM, Pereira AL, Ribeiro NF, Lino MMA, Dias LB, de Oliveira MFD, de Araujo-Silva OM, Dorneles MP, Vanin AA, Baroni BM, Bjordal JM, Casalechi HL, Leal-Junior ECP. Effects of photobiomodulation therapy combined with static magnetic field on training adaptations and detraining responses: a randomised placebo-controlled trial. BMJ Open Sport Exerc Med. 2025 Dec 12;11(4):e002799. doi: 10.1136/bmjsem-2025-002799. eCollection 2025. PMID 41393334
- [Derived] de Paiva PRV, Casalechi HL, Tomazoni SS, Machado CDSM, Vanin AA, Baroni BM, de Carvalho PTC, Leal-Junior ECP. Effects of photobiomodulation therapy combined to static magnetic field in strength training and detraining in humans: protocol for a randomised placebo-controlled trial. BMJ Open. 2019 Oct 28;9(10):e030194. doi: 10.1136/bmjopen-2019-030194. PMID 31662370